CLINICAL TRIAL: NCT02403388
Title: Implementation and Assessment of a Multifaceted Risk Management Program in French Multiprofessional Offices in Primary Care : the PRisM Study
Brief Title: Assessment of a Multifaceted Risk Management Program in French Multiprofessional Offices in Primary Care
Acronym: PRisM
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL14_0265
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2019-09

CONDITIONS: Risk Management; Primary Health Care; Patient Safety
Keywords: Patient safety; Primary care; Incident reporting; Pluridisciplinary care offices; Risk management; Assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Multiprofessional primary care offices with PRisM: 25 multiprofessional primary care offices. Each professional of care of the offices (about 10 FTE / office) have to declare each adverse event that occurs in their office during 18 months.
  Interventions: Other: PRisM
- Multiprofessional primary care offices without PRisM: 25 multiprofessional primary care offices. Each professional of care of the offices (about 10 FTE / office) have to declare each adverse event that occurs in their office during 18 months.

INTERVENTIONS:
Other: PRisM — A risk management program for each professional of care in multiprofessional primary care offices in France.
  Groups: Multiprofessional primary care offices with PRisM

SUMMARY:
Avoidable care associated incidents are relatively frequent in primary care. In France for example, avoidable incidents rate is estimated to 22/1000 medical acts from general practitioners. Patient safety is now a growing issue in primary care. One tool to increase patient safety is incident reporting and analysis. It could reduce some important consequences for patients and could allow implementing substantial corrective actions.

The aim of the PRisM study is to assess and compare the efficiency of a multifaceted risk management program implemented in the french pluridisciplinary offices in primary care in association with a centralized incident reporting system, versus a centralized incident reporting system only.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary multiprofessional primary care offices
* With at least 10 Full Time Equivalent (FTE)
* With at least general practitioners and 3 different occupations in care

Exclusion Criteria:

* Monoprofessional primary care offices

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Multiprofessional primary care offices in France (MSP, SS, PS)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2018-04-09 (Actual)

PRIMARY OUTCOMES:
Annual incident declaration rate by full-time equivalent in both groups. | 18 months

SECONDARY OUTCOMES:
Declaration rate of incident associated with patient injury in both groups | 18 months
Repartition of patient injury in different classes in both groups. | 18 months
Repartition of incidents causes in different classes in both groups. | 18 months
Repartition of preventive actions in different classes in both groups. | 18 months
Repartition of correctives actions in different classes in both groups. | 18 months
A mean score of french version of Medical Office Survey on Patient Safety (MOSPS) in both groups, including a mean score for each dimension of the survey. | 1 &18 months
Identification of brakes and levers (qualitative assessment) of program implementation in intervention group. | after 18 months
Psychometric analysis of Medical Office Survey on Patient Safety (french translation) for dimensional structuration of the survey. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Marc CHANELIERE, MD, Principal Investigator — Hospices Civils de Lyon, Pôle Information Médicale Evaluation Recherche
Locations (1):
- Pôle IMER - Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Derived] Chaneliere M, Buchet-Poyau K, Keriel-Gascou M, Rabilloud M, Colin C, Langlois-Jacques C, Touzet S. A multifaceted risk management program to improve the reporting rate of patient safety incidents in primary care: a cluster-randomised controlled trial. BMC Prim Care. 2024 Jul 6;25(1):244. doi: 10.1186/s12875-024-02476-4. PMID 38971743